CLINICAL TRIAL: NCT07364500
Title: Early Detection and Prevention of Health Complications in Premature Infants - Protocol-driven Nutrition
Brief Title: Protocol-driven Nutrition in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: General University Hospital, Prague (Other); University Hospital Olomouc (Other); České Budějovice Hospital (Other); Tomáš Baťa Regional Hospital in Zlín (Unknown); Brno University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UZIS 2025/2
Record Dates: First submitted 2026-01-13; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Preterm Infants
Keywords: preterm infants; nutrition of preterm infants; human milk analysis; nutrition monitoring; Czech Republic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preterm infants (Other): The nutritional management of enrolled patients will be guided by individualized plans developed by attending physicians, supported by advanced clinical nutrition software enabling precise monitoring and adjustment based on ongoing anthropometric and dietary data.
  Interventions: Dietary Supplement: Nutrition plan supported by advanced clinical nutrition software

INTERVENTIONS:
Dietary Supplement: Nutrition plan supported by advanced clinical nutrition software — Infants undergo regular anthropometric assessments (weight, length, head circumference), and detailed fluid and nutrient intake is recorded. Weekly analysis of the macronutrient composition of maternal or donor milk is conducted, enabling personalized fortification to meet the infant's current needs. The intervention utilizes a dedicated nutrition software tool, incorporating Fenton growth charts, to support clinical decisions and track progress via z-scores compared to term-born infants.
  By aligning nutrient supply with individual requirements and promoting early enteral feeding, the project seeks to enhance growth outcomes, minimize risks such as bronchopulmonary dysplasia or retinopathy, and shorten the length of stay in neonatal intensive care.

SUMMARY:
The project is a national, prospective, multicenter, interventional pilot project focused on protocol-driven nutrition in preterm infants in the Czech republic.

The primary aim of the project is to prepare, test, and develop a proposal for a national methodology for the care of preterm newborns in the field of nutrition. This will reduce health risks in premature infants and minimize the negative impacts on the overall development of the child and the family of the premature infant.

DETAILED DESCRIPTION:
The project is a national, prospective, multicenter, interventional pilot project focused on protocol-driven nutrition in preterm infants in the Czech republic.

The main goal of the project is standardization of nutrition of premature newborns across healthcare facilities with the aim to optimize postnatal growth and reduce complications associated with prematurity through individualized and closely monitored nutritional plans.

The project will be running in 5 perinatology centers in the Czech Republic. It is expected that 400 premature infants will participate. The project is supported by the European Social Fund (Operational Program Employment Plus) and the state budget of the Czech Republic and is registered by the Ministry of Labour and Social Affairs of the Czech Republic under ID: CZ.03.02.02/00/22_005/0002020. The study has been reviewed and approved by multiple local ethical committees. The listed IRB represents the lead national ethical committee overseeing the trial.

ELIGIBILITY:
Inclusion Criteria:

* Infants born before 31+6 weeks gestation.
* Signed consent for participation in the project and consent for the processing of personal data.
* Admission to neonatal care in the participating hospital within 24 hours after birth.

Exclusion Criteria:

* Congenital malformations.
* Fetal hydrops.
* Intraventricular hemorrhage requiring drainage.
* Necrotizing enterocolitis requiring surgical treatment.
* Surgically treated hydrocephalus.
* Unsigned consent for participation in the project and/or consent for the processing of personal data.

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Z-score for body weight at 36 weeks corrected gestational age | Up to a corrected gestational age of 36 weeks
Z-score for body length at 36 weeks corrected gestational age | Up to a corrected gestational age of 36 weeks
Z-score for head circumference at 36 weeks corrected gestational age | Up to a corrected gestational age of 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Plavka, prof., Study Director — General Hospital University in Prague; Jiří Dušek, M.D., MHA, Study Chair — České Budějovice Hospital
Locations (5):
- Czechia (5):
  - Brno University Hospital, Brno, Czech Republic
  - České Budějovice Hospital, České Budějovice, Czech Republic
  - University Hospital Olomouc, Olomouc, Czech Republic
  - General University Hospital, Prague, Czech Republic
  - Tomáš Baťa Regional Hospital in Zlín, Zlín